CLINICAL TRIAL: NCT04029610
Title: Evaluation of Cardiac Arrhythmias in Hand Surgery Using Local Anesthesia With Adrenaline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uri farkash (Other)
Responsible Party: Sponsor-Investigator, Uri farkash, Head, Hand Surgery Unit, Assuta Ashdod University Hospital, Assuta Ashdod Hospital
Organization: Assuta Ashdod Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 0002-17-AAA
Record Dates: First submitted 2019-07-20; First posted 2019-07-23 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Evaluation of Cardiac Arrhythmias in Hand Surgery Using Local Anesthesia With Adrenaline
MeSH Terms: interventions — Anesthesia, Local; Lidocaine; Epinephrine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Local anesthesia of lidocaine and arterial blockage on the arm (Active Comparator): Local anesthesia of lidocaine and arterial blockage on the arm
  Interventions: Drug: lidocaine and arterial blockage
- Local anesthesia with lidocaine and adrenalin (Experimental): Local anesthesia with lidocaine and adrenalin
  Interventions: Procedure: Local anesthesia with lidocaine and adrenalin.; Drug: lidocaine and adrenalin

INTERVENTIONS:
Procedure: Local anesthesia with lidocaine and adrenalin. — Local anesthesia with lidocaine and adrenalin.
  Arms: Local anesthesia with lidocaine and adrenalin
Drug: lidocaine and adrenalin — lidocaine and adrenalin
  Arms: Local anesthesia with lidocaine and adrenalin
Drug: lidocaine and arterial blockage — lidocaine and arterial blockage
  Arms: Local anesthesia of lidocaine and arterial blockage on the arm

SUMMARY:
Goals: 1. To check for frequency and type of arrhythmia in patients undergoing a medical procedure under local anesthesia 2. To examine whether the addition of adrenaline to local anesthesia affects the incidence of arrhythmias

DETAILED DESCRIPTION:
Rationale: Determining the frequency and type of arrhythmia will help determine the need for monitoring and the type of monitoring required during procedures under local anesthesia.

Patients will undergo the prescribed medical procedure using local anesthesia. Patients will be randomized into two groups: Group 1 - Local anesthesia of lidocaine and arterial blockage on the arm; Group 2 - Local anesthesia with lidocaine and adrenalin.

The amount and type of anesthetic used shall be recorded. In addition to the routine monitoring performed today (use of non-invasive blood pressure gauge and oxygen saturation), the patients will be connected to a cardiac holter monitor prior to the start of the surgical procedure and until they are released from the recovery room. Upon completion of the monitoring, the results of the holter test will be transmitted to the electrophysiology unit and analyzed to detect arrhythmias. There will be a registration of side effects reported by patients, which can result from arrhythmias (palpitations, dizziness, fainting, CPR). In patients in whom arrhythmias are detected, the type of arrhythmia and if it was accompanied by clinical symptoms will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who undergo hand surgery using local anesthesia at Assuta Ashdod Hospital

Exclusion Criteria:

* Patients with a known medical history of cardiac arrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Arrhythmia | 1 day of procedure
  Arrhythmia

CONTACTS AND LOCATIONS:
Overall Officials: Uri Farkash, MD, Principal Investigator — Head, Hand Surgery Unit, Assuta Ashdod Hospital
Locations (1):
- Assuta Ashdod Hospital, Ashdod, Israel

IPD SHARING:
Plan to Share IPD: No